CLINICAL TRIAL: NCT05219838
Title: Interventional , Open-label, Positron Emission Tomography (PET) Study With [18F]-T-401 Investigating MAGL Enzyme Occupancy After Multiple Oral Doses of Lu AG06466
Brief Title: Binding and Effects of Lu AG06466 in the Brain of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19941A
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AG06466 Low Dose (Experimental): Participants will receive Lu AG06466 low dose capsule orally once daily for 6 days approximately 30 minutes following a light meal.
  Interventions: Drug: Lu AG06466
- Lu AG06466 High Dose (Experimental): Participants will receive Lu AG06466 high dose capsule orally once daily for 6 days approximately 30 minutes following a light meal.
  Interventions: Drug: Lu AG06466

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 will be administered per dose and schedule specified in the arm description.

SUMMARY:
This study is being done to learn about the binding of Lu AG06466 and its major breakdown product (Lu AG06988) in the brain of healthy men having received multiple doses of Lu AG06466. As the binding will result in inhibition of an enzyme in the endocannabinoid system called monoacylglycerol lipase (MAGL), the effects on this system will be evaluated both in the blood and cerebrospinal fluid and compared to the binding in the brain.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18 and ≤30 kilograms (kg)/square meter (m^2) at the screening visit.
* The participant has a weight of ≥60 kg at the screening visit and baseline visit.
* The participant has a waist circumference ≤94 centimeters (cm) at the screening visit.

Exclusion Criteria:

* The participant has taken disallowed medication <2 weeks prior to the first dose of study drug or <5 half-lives prior to the screening visit for any medication taken.
* The participant has received a COVID-19 vaccination within the last 30 days before receiving first dose of study drug.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Lu AG06466 and Lu AG06988 | Day 5 (pre-dose, per hour before and after positron emission tomography [PET] imaging and per 30 minutes during PET imaging) and on Day 6 (3 hours post-dose)
Cerebrospinal Fluid (CSF) Concentration of Lu AG06466 and Lu AG06988 | Pre-dose and on Day 6 (3 hours post-dose)
Central MAGL Occupancy (%) Measured Using [18F]MNI-1188 PET Imaging | 2 to 4 hours post-dose on Day 5
CSF Concentrations of 2-arachidonolylglycerol (2-AG) (1-arachidonolylglycerol [1-AG]+2-AG), 2-oleoylglycerol (2-OG), and arachidonic acid (AA) | Day 6 (3 hours post-dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Invicro, LLC, New Haven, Connecticut, United States